CLINICAL TRIAL: NCT00816998
Title: The Effect of Early vs. Delayed Range of Motion in the Outcome of Patients With Distal Radius Fractures
Brief Title: Range of Motion and Patients With Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Alexander Y. Shin, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-004364
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Radius Fractures
Keywords: Radius fractures
MeSH Terms: conditions — Radius Fractures | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early (Other): Participants randomized to this arm will begin physical therapy of their fractured wrist approximately one week following surgery
  Interventions: Procedure: Physical therapy
- Delayed (Other): Participants randomized to this group will begin physical therapy of their fractured wrist approximately 6 weeks from their surgery. This is the approximate time frame in which therapy begins for patients not involved in the study. The term Delayed refers to therapy being delayed in starting from those in the study who begin therapy at one week post-operatively, not a delay in current care practice.
  Interventions: Procedure: Physical therapy

INTERVENTIONS:
Procedure: Physical therapy — Physical therapy to instruct participant with exercises to assist in return to normal activities following the healing of their wrist fracture
Procedure: Physical Therapy — Physical therapy to include exercises to help a participant improve the range of motion, grip and pinch strength following the fracture of their wrist

SUMMARY:
Hypothesis : Early active range of motion protocol after open reduction and internal fixation of a distal radius fracture with a volar fixed angle locking plate results in earlier return of functional motion, earlier return to work and improved functional outcomes compared delayed mobilization.

Specific Aim:

To compare early range of motion versus delayed motion protocol in distal radius fractures treated with open reduction and internal fixation with a volar fixed angle locking plate with respect to time to fracture union, range of motion, functional outcome measures, return to work and complications.

DETAILED DESCRIPTION:
You are scheduled for surgery of your broken wrist. Treatment of broken bones of the wrist, such as distal radius fractures, may require different types of treatment. For this study this type of fracture will be treated by surgery to place a plate with screws to the broken bone and then a plaster splint will be applied. After surgery, physical therapy will be started. Following surgery you will be assigned to one of four groups by the type of wrist fracture (broken bone) you have. Each person will by chance (the flip of a coin) be put in either the Early or Delayed Range of Motion groups. Those in the Early Range of Motion groups will begin exercises for motion starting 7 days after surgery. Those in the Delayed Range of Motion, will begin exercises for motion starting about five weeks after surgery. Once you begin the exercises to help you get back normal use of your wrist, you will have measurements of how much motion and strength you have in the wrist and hand that was fractured. The measurements will take about five minutes to complete. All participants will have an x-ray of the wrist at 2, & 6 weeks following surgery and if needed at other appointments. At each appointment you will be asked to fill out four questionnaires, asking about pain and how you are getting along with the broken bone in your wrist. The questionnaires will take about 20 minutes of your time to complete. At Week 26 you will be asked to record the amount of motion you have in both of your wrists on paper drawings as well as the measurements that we will make. Working with the drawings will take approximately five minutes. At Week 52 you will be asked two questions about how satisfied you are with the results of your surgery. Surgery, x-ray of your wrist, and exercise to help you get back motion of your broken wrist are all standard orthopedic practice for treating a broken wrist bone.

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be met to be enrolled:

1. Have a closed unstable distal radius fracture
2. Have a fracture classified as an AO Type A or C fracture, with or without an ulnar styloid fracture
3. Be a male or non-pregnant female at least 18 years of age.
4. Understand the requirements of the study and able to provide a written informed consent and comply with the study protocol
5. Have the ability to understand and provide written authorization for use and disclosure of personal health information

Exclusion Criteria:

Participants are excluded if they:

1. Have any of the following conditions

   1. Concomitant contralateral or ipsilateral upper extremity fractures
   2. Ipsilateral ulna (excluding styloid) fracture
   3. Open, multi-fragmentary fracture
   4. Artery or Nerve injury secondary to fracture
2. Have had a previous ipsilateral distal radius fracture in the 2 years prior to enrollment
3. Are currently on chemotherapy or radiation therapy
4. A history of a metabolic disorder affecting the skeletal system other than osteoarthritis or osteoporosis
5. A history of uncontrolled diabetes
6. Are unable to provide consent for the study
7. Are unable to make the follow-up appointments required of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Range of motion measurements | at each study visit

SECONDARY OUTCOMES:
Pinch strength | at each study visit
Grip strength | at each study visit
Pain | at each study visit
Return to work | at each study visit
Scores of DASH & PRWE questionnaires | at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Y. Shin, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States